CLINICAL TRIAL: NCT00808691
Title: Microcirculation and Oxidative Stress in Critically Ill Patients in Surgical Intensive Care Unit
Brief Title: Microcirculation and Oxidative Stress in Critical Ill Patients in Surgical Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200707012
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Sepsis; ARDS; Liver Failure; Renal Failure; Brain Death
MeSH Terms: conditions — Sepsis; Liver Failure; Renal Insufficiency; Brain Death | interventions — Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: Patients with sepsis
  Interventions: Other: Critical care
- 2: Patient admitted for postoperative care
  Interventions: Other: Critical care
- 3: Patients with ARDS
  Interventions: Other: Critical care
- 4: Patients with ARF
  Interventions: Other: Critical care
- 5: Patients who receive liver support treatment
  Interventions: Other: Critical care
- 6: Patients wiht brain death
  Interventions: Other: Critical care

INTERVENTIONS:
Other: Critical care — Standard care for each group of patients

SUMMARY:
As medicine advances, many lives can be saved in the intensive care unit. However, when multiple organ failure occurs, the mortality rate of patients increases dramatically. Therefore, the major goal in the intensive care unit is to prevent the occurrence of multiple organ failure. The sepsis protocol and early goal directed treatment have great effects to reduce development of multiple organ failure and to decrease the mortality rate. However, sometime the condition of patient deteriorated in spite of both the mean blood pressure and mixed venous oxygen saturation are normal. Some experts recognize that there might be microcirculatory dysfunction of tissue or organ. The dysfunction of microcirculation might due to vasoconstriction or microthrombosis. Vasoconstriction might result from systemic inflammation, reactive oxygen species, or dysfunction of synthesis of NO (nitric oxide). Microthrombosis might result from systemic inflammation, reactive oxygen species, imbalance of coagulatory system, or damage of endothelial cell.

In clinical practice, the oxidative stress is related to circulatory shock, sepsis, acute lung injury, and acute respiratory distress syndrome. This study tries to investigate the relation between oxidative stress and microcirculation. Furthermore, the investigators will try to investigate the correlation between the severity of oxidative stress and microcirculatory dysfunction and the severity of disease and prognosis. The investigators hope this study will help them to figure out the picture of disease progression of patients. It may conduct further study to modulate the oxidative stress, to improve the microcirculatory function, and finally to improve the outcome of patients.

ELIGIBILITY:
Inclusion Criteria:

* > 18 y/o
* Related diagnosis made within 24h
* Group 1 - Sepsis
* Group 2 - Postoperative care
* Group 3 - ARDS
* Group 4 - Renal failure
* Group 5 - Liver failure
* Group 6 - Brain death

Exclusion Criteria:

* Pregnant patients
* Related diagnosis made longer than 24h
* Patients who have received antioxidants within 24h
* Patients who have received hyperbaric oxygen therapy
* Patients who have a hemoglobin value less than 9 g/dl
* Patients who have received NO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paitents admitted to intensive care unit with the following conditions Sepsis Postoperative care ARDS Renal Failure Liver failure Brain death
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Mortality Severity of Organ Failure | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, M.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan